CLINICAL TRIAL: NCT00426998
Title: A 24 Month Randomized, Double-Masked, Single Center, Phase II Study Comparing Photodynamic Therapy With Verteporfin (Visudyne)Plus Two Different Timing Regimens of Intravitreal Bevacizumab (Avastin) Given 1 Week Prior to or 1 Week Following Photodynamic Therapy in Patients With Subfoveal Choroidal Neovascularization Secondary to Age-Related Macular Degeneration.
Brief Title: Combination Bevacizumab and Verteporfin (Two Different Sequences of Treatment)in Neovascular AMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Retinal Consultants Medical Group (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ComB-V001
Record Dates: First submitted 2007-01-24; First posted 2007-01-26 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Choroidal Neovascularization; Macular Degeneration
Keywords: Choroidal neovascularization due to age-related macular degeneration
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration | interventions — Verteporfin; Bevacizumab

INTERVENTIONS:
Drug: Verteporfin
Drug: Bevacizumab

SUMMARY:
The purpose of this research study is to compare different timing therapies of Verteporfin with Bevacizumab to treat choroidal neovascularization (CNV) due to age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

1. Patients are men or women of age 55 or older
2. Patients have subfoveal CNV due to AMD with lesion size less than or equal to 9 MPS DA
3. patients have not received previous treatment for subfoveal CNV due to AMD.
4. Patients have a visual acuity between 20/40 and 20/320-

Exclusion Criteria:

1. Subjects who have received previous treatment for subfoveal CNV, in their study eye including prior PDT, transpupillary thermotherapy (TTT), submacular surgery, drug therapies such as Macugen or other anti-angiogenic compounds, or other local treatment. Previous laser photocoagulation therapy is acceptable, provided it was not subfoveal.
2. Patients with a known hypersensitivity/allergy to verteporfin, porfimer sodium, or other porphyrins, porphyria or other porphyrin sensitivity, or hypersensitivity to sunlight or bright artificial light.
3. Patients who use medications that may induce photosensitivity.
4. Patients who have undergone YAG capsulotomy within the last month.
5. Subjects currently involved in any experimental procedure within the last 12 weeks.
6. Female patients who are pregnant, fecund or breast-feeding.

   -

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-04

PRIMARY OUTCOMES:
percentage of patients losing 3 or more lines of visual acuity
percentage of patients gaining 3 or more lines of visual acuity
mean change from baseline in visual acuity
OCT evidence of active CNV leakage
fluorescein angiographic evidence of active CNV leakage
number of retreatments

CONTACTS AND LOCATIONS:
Overall Officials: Joel A Pearlman, M.D., Ph. D., Principal Investigator — Retinal Consultants Medical Group, Inc.
Locations (1):
- Retinal Consultants Medical Group, Inc., Sacramento, California, United States